CLINICAL TRIAL: NCT06820788
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effect of Music on Pain and Comfort Levels After Laparoscopic Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: okutan6
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Surgery
Keywords: music therapy; pain; laparoscopic surgery; comfort
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-testpost-test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): As part of the pre-test, the patient introduction form, comfort and pain scales will be applied to the experimental group patients. Music will be played in the patient room 2 hours after the patients are transferred from the post-operative care unit to the clinic, which is the most appropriate time after surgery, when vital signs are stable and clinical compliance is achieved. Music will be played for 20 minutes. As part of the post-test, the comfort and pain scales will be applied to the experimental group patients again.
  Interventions: Other: music therapy
- Control Group (No Intervention): As part of the pre-test, the patient introduction form, comfort and pain scales will be applied to the control group patients. No intervention will be applied to the control group patients and the clinic's routine practices will continue. As part of the post-test, the comfort and pain scales will be applied to the control group patients again.

INTERVENTIONS:
Other: music therapy — Local music will be played in the patient room 2 hours after the patient is transferred from the postoperative care unit to the clinic, which is the most appropriate time after surgery, when vital signs have stabilized and clinical adaptation has been achieved.
  Arms: Intervention Group

SUMMARY:
It is planned to examine the effects of local music on pain and comfort levels in patients undergoing laparoscopic abdominal surgery and to make a comparison between Turkey and Iran with the results obtained.

The hypotheses of the study are as follows:

H1-0: Music has no effect on reducing pain in patients undergoing laparoscopic abdominal surgery.

H1-1: Music has an effect on reducing pain in patients undergoing laparoscopic abdominal surgery.

H2-0: Music has no effect on increasing comfort in patients undergoing laparoscopic abdominal surgery.

H2-1: Music has an effect on increasing comfort in patients undergoing laparoscopic abdominal surgery.

DETAILED DESCRIPTION:
As part of the pre-test, the patient introduction form, comfort and pain scales will be applied to the experimental group patients. Music will be played in the patient room 2 hours after the patients are transferred from the post-operative care unit to the clinic, which is the most appropriate time after surgery, when vital signs are stable and clinical compliance is achieved. Music will be played for 20 minutes. As part of the post-test, the comfort and pain scales will be applied to the experimental group patients again.

As part of the pre-test, the patient introduction form, comfort and pain scales will be applied to the control group patients. No intervention will be applied to the control group patients and the clinic's routine practices will continue. As part of the post-test, the comfort and pain scales will be applied to the control group patients again.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years old
* Must not have communication problems

Exclusion Criteria:

* Having any hearing or mental problems
* Laparoscopic surgery converted to open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
pain level | The patients will be given the scale in the patient room 2 hours after the surgery. The scale will be given again as a final test immediately after the music listening is over.
  Numerical Rating Scale:
  This scale, which is intended to determine the severity of pain, aims to have the patient describe their pain with numbers. In the form, 0 points are evaluated as "no pain", 1-3 points as "mild pain", 4-6 points as "moderate pain", and 7 and above points as "severe pain"
comfort level | The patients will be given the scale in the patient room 2 hours after the surgery. The scale will be given again as a final test immediately after the music listening is over.
  General Comfort Scale Short Form:
  General Comfort Scale Short Form is the Turkish adaptation of the General Comfort Scale developed by Kolcaba to measure the individual's comfort level in a more understandable way and in a shorter time. The scale consists of 28 items and the items of the scale are scored between 28-168. High scores indicate a high level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)